CLINICAL TRIAL: NCT03346512
Title: Considerations on the Transfusion Threshold in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-perfusion
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery: Patients having undergone cardiac surgery (other than the placement of a pacemaker or defibrillator) within the CHU Brugmann hospital between 2006 and 2015
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Cardiac surgery

SUMMARY:
This is a retrospective observational study of the transfusion threshold in cardiac surgery.

There is controversy in the literature regarding the transfusion threshold to be adopted, especially in a patient who has undergone cardiac surgery. Some authors suggest that the transfusion should be done in a restrictive way when a certain threshold in hemoglobin is reached, in order to avoid the risks it implies, especially infectious.This threshold is very controversial and remains to be defined (variations in the literature from 7g / dL to 9g / dL). Other authors conclude that there is no superiority of a restrictive transfusion compared to a more liberal transfusion, with regard to the morbidity or medical costs.

It is therefore interesting to study, in a retrospective manner, the global and multidisciplinary management of patients who have undergone a cardiac surgery within the CHU Brugmann hospital, to analyze if they have been adequately transfused.

ELIGIBILITY:
Inclusion Criteria:

- Patients having undergone cardiac surgery (other than the placement of a pacemaker or defibrillator) within the CHU Brugmann hospital between 2006 and 2015

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having undergone cardiac surgery (other than the placement of a pacemaker or defibrillator) within the CHU Brugmann hospital between 2006 and 2015
Sampling Method: Non-Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

PRIMARY OUTCOMES:
Hemoglobin rate | Baseline (just before cardiac surgery)
  Hemoglobin rate
Hemoglobin rate | One day after surgery (J1)
  Hemoglobin rate
Hemoglobin rate | Two days after surgery (J2)
  Hemoglobin rate
Hemoglobin rate | Five days after surgery (J5)
  Hemoglobin rate
Hematocrit rate | Baseline (just before cardiac surgery)
  Hematocrit rate
Hematocrit rate | One day after surgery (J1)
  Hematocrit rate
Hematocrit rate | Two days after surgery (J2)
  Hematocrit rate
Hematocrit rate | Five days after surgery (J5)
  Hematocrit rate
International Normalized Ratio (INR) | Baseline (just before cardiac surgery)
  Coagulation indicator
International Normalized Ratio (INR) | One day after surgery (J1)
  Coagulation indicator
International Normalized Ratio (INR) | Two days after surgery (J2)
  Coagulation indicator
International Normalized Ratio (INR) | Five days after surgery (J5)
  Coagulation indicator
Creatinin rate | Baseline (just before cardiac surgery)
  Renal function indicator
Creatinin rate | One day after surgery (J1)
  Renal function indicator
Creatinin rate | Two days after surgery (J2)
  Renal function indicator
Creatinin rate | Five days after surgery (J5)
  Renal function indicator
Total amount of blood perfusions | Five days after surgery (J5)
  Total amount of blood perfusions
Liquid balance | One day after surgery
  Ratio between total fluid intake (perfusion) and loss (blood and urine)

CONTACTS AND LOCATIONS:
Overall Officials: Kenza Bradly, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No